CLINICAL TRIAL: NCT01421550
Title: Conservative Treatment Versus Elective Repair of the Umbilical Hernia in Patients With Ascites and Liver Cirrhosis, a Randomized Controlled Trial
Brief Title: Conservative Treatment Versus Elective Repair of Umbilical Hernia in Patients With Ascites and Liver Cirrhosis
Acronym: CRUCIAL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, hasan eker, Dr. G. Kazemier, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRUCIAL trial
Record Dates: First submitted 2011-08-19; First posted 2011-08-23 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Umbilical Hernia; Liver Cirrhosis; Ascites
Keywords: umbilical; hernia; cirrhosis; ascites; conservative; surgery; optimal management
MeSH Terms: conditions — Hernia, Umbilical; Liver Cirrhosis; Ascites; Hernia; Fibrosis | interventions — Conservative Treatment; Wound Healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conservative treatment (Active Comparator): Patients that randomize for conservative management of their umbilical hernia will be followed routinely at the polyclinical ward.
  Interventions: Procedure: Conservative treatment
- Surgical repair (Active Comparator): Patients that randomize for surgical repair of their umbilical hernia will be operated in an elective setting after a careful preoperative work-up.
  Interventions: Procedure: Surgical repair

INTERVENTIONS:
Procedure: Conservative treatment — Patients that randomize for conservative management of their umbilical hernia will be followed routinely at the polyclinical ward.
  Arms: Conservative treatment
Procedure: Surgical repair — Patients that randomize for surgical repair of their umbilical hernia will be operated in an elective setting after a careful preoperative work-up.
  Arms: Surgical repair

SUMMARY:
The purpose of the present study is to investigate whether or not to perform elective surgical repair of umbilical hernias in patients with liver cirrhosis and ascites. There are no other randomized controlled trials in this area. The optimal management in patients with umbilical hernias and liver cirrhosis with ascites is not clear yet. The general surgical opinion is that umbilical hernias in patients with ascites should not be corrected because of the supposedly high operative risks and high recurrence rates. Conservative treatment, however, can have severe complications resulting in emergency repair. Such operations carry a higher risk of complications than elective operations, particularly in this group of patients. Prospective and retrospective series showed us that elective hernia repair in this specific patient group is safe without major complications or high recurrence rates.

The aim of this study is to asses the optimal timing of correction of umbilical hernia in patients with liver cirrhosis and ascites.

ELIGIBILITY:
Inclusion Criteria:

* Primary Umbilical hernia
* Liver cirrhosis
* Ascites (US proven)
* Age ≥ 18 years
* Signed Informed consent

Exclusion Criteria:

* Recurrent umbilical hernia
* Midline laparotomy in medical history
* ASA1 score IV or above
* Incarcerated hernia related emergency procedures
* Patent umbilical vein; >5mm
* Expected time to Ltx <3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
complications | 2 years
  The primary endpoint in this study is a composite endpoint of the overall morbidity after 24 months, which includes; Reoperation for complication (e.g. hemorrhage; Decompensated liver failure(e.g. Portal vein thrombosis; Non-closure of surgical wound at 4 weeks; Haematoma; Seroma; Rupture of hernia; Bowel incarceration; Necrosis and rupture of the overlying skin; Evisceration; Pneumonia; Urinal tract infection; Postoperative surgical site infection (superficial/deep/organ space); Postoperative leakage of ascites more than 2 weeks after surgery

SECONDARY OUTCOMES:
Recurrence | 2 years
Mortality | 2 years
Length of hospital stay | 3 months
Quality of life | 2 years
Cost effectiveness | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: G Kazemier, MD, PhD, Principal Investigator — Erasmus Medical Center; J.F. Lange, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Derived] de Goede B, van Rooijen MMJ, van Kempen BJH, Polak WG, de Man RA, Taimr P, Lange JF, Metselaar HJ, Kazemier G. Conservative treatment versus elective repair of umbilical hernia in patients with liver cirrhosis and ascites: results of a randomized controlled trial (CRUCIAL trial). Langenbecks Arch Surg. 2021 Feb;406(1):219-225. doi: 10.1007/s00423-020-02033-4. Epub 2020 Nov 25. PMID 33237442